CLINICAL TRIAL: NCT01145053
Title: Long Time Survey of RESPIMAT in Daily Clinical Use
Brief Title: Drug Use Survey of RESPIMAT in Patients With COPD
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.463
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Results first posted 2013-01-30 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Treatment

SUMMARY:
To investigate safety and effectiveness information on the use of Tiotropium Respimat for long time of period in daily practical clinical circumstances, and to obtain proper drug use information.

ELIGIBILITY:
Inclusion criteria:

Patients with COPD who is expected to be treatable with long term. All patients must have a diagnosis of COPD and register after the start of treatment of Tiotropium Respimat.

Exclusion criteria:

There is no special restriction, because this PMS is an observational investigation under conditions of normal clinical practice. Spiriva Respimat is contraindicated in patients with hypersensitivity to Tiotropium bromide, atropine or its derivatives, e.g. ipratropium or oxitropium or to any of the excipients in Package labelling.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 300
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 361 patients were enrolled. Of these patients, the CRF of 4 patients were uncollected by reason of institution, and the 16 patients who did not visit after enrollment. Then, total 341 patients were observed in the survey.
Groups:
- Spiriva Respimat: Spiriva 2.5 mcg Respimat 60 puffs
Period: Overall Study
Arm/Group | Spiriva Respimat
Started | 341
Completed | 248
Not Completed | 93
Not completed — Adverse Event | 22
Not completed — Lost to Follow-up | 28
Not completed — Withdrawal by Subject | 25
Not completed — Other | 18

BASELINE CHARACTERISTICS:
Arm/Group | Spiriva Respimat
Number analyzed (Participants) | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 294

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events (AEs)
Description: The number of patient with any AEs, patients with drug-related AEs
Time Frame: Week 52
Population: The all treated patients
Measure: Number; unit: Patients
Arm/Group | Spiriva Respimat
Number analyzed (Participants) | 341
Patients
  patient with any AEs | 53
  patients with drug-related AEs | 16

2. Secondary Outcome: Effectiveness
Description: Effectiveness should be comprehensively investigated based on the items of patients observation, test results of FEV1, clinical symptoms. The Effectiveness is classified into 3 category, 'Improved', 'No change' and 'Aggravated' by physician.
Time Frame: Week 52
Population: The 25 patients which were non approved indication patients and no efficacy information, were excluding from safety set, 316 patients were included in efficacy set.
Measure: Number; unit: Patients
Arm/Group | Spiriva Respimat
Number analyzed (Participants) | 316
Patients
  Improved | 191
  No change | 122
  Aggravated | 3

3. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1)
Description: FEV1 is observed at Week 0 and Week 52. The change of FEV1 from Week 0 to Week 52 is calculated.
Time Frame: Week 0 and Week 52
Population: The 25 patients which were non approved indication patients and no efficacy information, were excluding from safety set, 316 patients were included in efficacy set. In the efficacy set, 105 patients measured FEV1 .
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Spiriva Respimat
Number analyzed (Participants) | 105
L
  Week 0 | 1.39 (0.66)
  Week 52 | 1.46 (0.66)
  Change from Week 0 to Week 52 | 0.06 (0.28)

4. Secondary Outcome: Cough Frequency
Description: Cough frequency is rating 1 to 4 score based on patient's diary: 1=None; 2=A few times; 3=Frequently; 4=Very frequently.
Time Frame: Week 0 and Week 52
Population: The 25 patients which were non approved indication patients and no efficacy information, were excluding from safety set, 316 patients were included in efficacy set. In the efficacy set, 309 patients recorded the Cough Frequency .
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Spiriva Respimat
Number analyzed (Participants) | 309
Units on a scale
  Week 0 | 2.10 (0.69)
  Week 52 | 1.62 (0.59)
  Change from Week 0 to Week 52 | -0.47 (0.63)

5. Secondary Outcome: Amount of Sputum
Description: Amount of Sputum is rating 1 to 4 score based on patient's diary: 1= None; 2= Slight; 3=Slightly more; 4= Very much.
Time Frame: Week 0 and Week 52
Population: The 25 patients which were non approved indication patients and no efficacy information, were excluding from safety set, 316 patients were included in efficacy set. In the efficacy set, 309 patients recorded the Amount of Sputum.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Spiriva Respimat
Number analyzed (Participants) | 309
Units on a scale
  Week 0 | 2.05 (0.74)
  Week 52 | 1.63 (0.61)
  Change from Week 0 to Week 52 | -0.42 (0.63)

6. Secondary Outcome: Shortness of Breath
Description: Shortness of Breath is rating 1 to 6 score based on patient's diary: 1=No shortness of breath and no problem in activity in daily life (ADL); 2=Despite shortness of breath, can move about like other people of the same age and no problem in ADL; 3=Can walk fast for a short time but activities like other people of the same age are not possible; 4=Can walk normally, go up the stairs slowly but quick motion is difficult; 5=Can walk slowly in the neighborhood but shortness of breath occurs; 6= Due to severe shortness of breath, rested at home all day.
Time Frame: Week 0 and Week 52
Population: The 25 patients which were non approved indication patients and no efficacy information, were excluding from safety set, 316 patients were included in efficacy set. In the efficacy set, 309 patients recorded the Shortness of Breath.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Spiriva Respimat
Number analyzed (Participants) | 309
Units on a scale
  Week 0 | 3.28 (1.29)
  Week 52 | 2.69 (1.34)
  Change from Week 0 to Week 52 | -0.59 (0.82)

7. Secondary Outcome: Nocturnal Sleep
Description: Nocturnal Sleep is rating 1 to 5 score based on patient's diary: 1=Sputum and cough hardly made me awake; 2=Sputum and cough only one time made me awake; 3=Sputum and cough 2 or 3 times made me awake; 4=Sputum and cough 4 to 6 times made me awake; 5=Sputum and cough made me awake all night.
Time Frame: Week 0 and Week 52
Population: The 25 patients which were non approved indication patients and no efficacy information, were excluding from safety set, 316 patients were included in efficacy set. In the efficacy set, 308 patients recorded the Nocturnal Sleep.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Spiriva Respimat
Number analyzed (Participants) | 308
Units on a scale
  Week 0 | 1.55 (0.84)
  Week 52 | 1.25 (0.60)
  Change from Week 0 to Week 52 | -0.31 (0.58)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Spiriva Respimat
Serious Adverse Events (participants affected / at risk) | 27/341
Other Adverse Events (participants affected / at risk) | 0/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiriva Respimat (N=341)
Cardiac failure (Cardiac disorders) | 1
Cor pulmonale (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Maculopathy (Eye disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Pneumonia (Infections and infestations) | 4
Pneumonia bacterial (Infections and infestations) | 3
Atypical mycobacterial infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Loss of consciousness (Nervous system disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes